CLINICAL TRIAL: NCT05583266
Title: Efficacy of Pentoxifylline on Cerebrovascular Function in Patients With Cerebral Small Vessel Disease(PERFORM)：A Randomized, Double-blinded, Placebo-controlled, Multi-center Trial
Brief Title: Efficacy of Pentoxifylline on Cerebrovascular Function in Patients With Cerebral Small Vessel Disease(PERFORM)
Acronym: PERFORM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, yilong Wang, Vice President of Beijing Tiantan Hospital, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KY2022-100-02
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: cerebral small vessel diseases; Pentoxifylline; randomized controlled trial; multicenter study; double blind study; placebo-controlled
MeSH Terms: conditions — Cerebral Small Vessel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pentoxifylline sustained- release tablets placebo group (Placebo Comparator): This group will receive Pentoxifylline sustained-release tablets placebo, 1 tablet twice a day, from the day of randomization to 6 months.
  Interventions: Drug: Pentoxifylline sustained-release tablets placebo
- Pentoxifylline sustained- release tablets group (Experimental): This group will receive Pentoxifylline sustained-release tablets, 1 tablet twice a day, from the day of randomization to 6 months.
  Interventions: Drug: Pentoxifylline sustained-release tablets

INTERVENTIONS:
Drug: Pentoxifylline sustained-release tablets — a dose of 1 tablet twice a day of Pentoxifylline sustained-release tablets
  Arms: Pentoxifylline sustained- release tablets group
Drug: Pentoxifylline sustained-release tablets placebo — Pentoxifylline sustained-release tablets placebo will be administrated at the same dosage and frequency as the experimental group
  Arms: Pentoxifylline sustained- release tablets placebo group

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, multi-center trial. Cerebral small vessel disease (CSVD) patients will be diagnosed according to STRIVE standards and randomized into the Pentoxifylline sustained-release tablet group and placebo group. The purpose of this trial is to assess the efficacy of Pentoxifylline sustained- release tablets on CSVD.

DETAILED DESCRIPTION:
Cerebral small vessel disease (CSVD) is a complex whole brain disease, which is a series of clinical, imaging, and pathological syndromes caused by various etiologies affecting small arteries, micro-arteries, capillaries, micro-venules, and small veins in the brain, and is a common clinical vascular disease of the brain, usually with insidious onset, slow progression, and some acute attacks.

The incidence of CSVD is positively correlated with age. Studies have shown that in people aged 60 to 70 years, 87% had subcortical white matter lesions and 68% had periventricular white matter changes, whereas, in people aged 80 to 90 years, 100% had subcortical white matter changes and 95% had periventricular changes. The incidence of cerebral microhemorrhage is approximately 6% in the 45-50 years old population and up to 36% in the 80-year-old population.

Pentoxifylline, a xanthine derivative, is mainly used for the improvement of cerebral circulation after ischemic cerebrovascular disease and for peripheral vascular disease, such as chronic occlusive vasculitis with intermittent claudication treatment. Pentoxifylline is a non-selective phosphodiesterase inhibitor that increases intracellular cyclic AMP (cAMP) and activates protein kinase A31, playing an anti-inflammatory, anti-oxidation, inhibition of platelet aggregation, and vasodilation. Pentoxifylline is a well-tolerated drug for improving peripheral blood flow disorders, primarily by increasing blood flow and increasing oxygenation of ischaemic tissues. In addition, it improves vasodilatation by increasing prostacyclin and has a specific effect on the immune response by inhibiting tumor necrosis factors.

Patients meeting the enrollment criteria will be randomly assigned to one of the two treatment groups with the use of a double-blind design (a dose of 1 tablet twice a day, from randomization to 6 months). Face-to-face interviews will be conducted at baseline, on day 30 after randomization, on day 90 after randomization, and on day 180 after randomization.

The primary endpoint was the change in cerebral blood flow (CBF) and pulsatility index of the middle cerebral artery (MCA) after 6 months of treatment based on transcranial doppler (TCD) assessment of enrolled patients. The secondary endpoints include changes in clinical symptoms, MRI imaging markers (white matter hyperintensity, lacunes, microbleeds, enlarged perivascular space), and cognitive function at 6 months. The safety endpoints include moderate or severe hemorrhage events, symptomatic and asymptomatic intracranial hemorrhage, overall mortality, and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Age 45-75 years;
2. CSVD can be seen on MRI, which satisfies one of the following conditions:

   * Presence of white matter hyperintensities and Fazekas score ≥2;
   * Lacunar Infarction ≥1, with or without white matter hyperintensities;
3. is eligible for Transcranial Doppler (TCD) monitoring;
4. meeting the following clinical manifestations:

   * Patients with vascular cognitive impairment (abnormalities in memory and or other cognitive domains lasting at least 3 months) ;
   * MoCA ≤22 points; MoCA ≤21 points for primary education and below;
5. independent in daily life (modified mRS ≤2) ;
6. with signed informed consent.

Exclusion Criteria:

1. patients with acute cerebral infarction and acute cerebral hemorrhage;
2. patients with bleeding tendency: including platelet count < 100 × 10*9/L, active peptic ulcer, history of intracranial hemorrhage (such as epidural hematoma, subdural haematoma, subarachnoid hemorrhage, cerebral hemorrhage, etc.) , cerebral microbleedings (≥5 cerebral microbleedings) , brain tumor, cancer-related stroke, taking anticoagulant drugs, or using dual antiplatelet therapy;
3. patients who have a history of cognitive impairment caused by other causes, such as normal pressure hydrocephalus, Alzheimer's disease, Parkinson's disease, multiple sclerosis, encephalitis, etc.;
4. patients with acute coronary syndrome and severe coronary arteriosclerosis;
5. patients with severe hepatic insufficiency, renal insufficiency, or severe cardiac insufficiency before randomization (severe hepatic insufficiency refers to ALT ≥2.0 times the upper limit of normal or AST ≥2.0 times the upper limit of normal; severe renal insufficiency refers to CRE ≥1.5 times the upper limit of normal or EGFR < 40 ml/min/1.73 m2; severe cardiac insufficiency refers to NYHA grade of 3-4) ;
6. patients who are pregnant, lactating or likely to become pregnant and planning to become pregnant;
7. patients with refractory hypertension;
8. patients with known allergic history to pentoxifylline, methylxanthine (such as caffeine, aminophylline, dihydroxypropyltheophylline, etc.) ;
9. patients with use of other vasodilators or circulatory improvers within 1 week (e.g. Cilostazol, Vinpocetine, Dimitamol, Sildenafil, Butylphthalide, Betahistine, Uracillin, Alprostadil, etc.) May stop taking the drug for 1 week before enrolling if criteria are met;
10. Patients using other drugs that affect the safety or efficacy evaluation of the tiral drug and who do not agree to discontinue the drug, such as GLP-1 receptor agonists, Liraglutide, dulasapeptide, risperidone, and exenatide;
11. Patients with other life-threatening or serious diseases with an expected survival of < 36 months;
12. Patients with contraindications to MRI;
13. Patients who could not cooperate to complete the follow-up;
14. Patients who enrolled in other clinical trials within 30 days.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2023-03-03 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
The change in cerebral blood flow at 6 months | 3 months and 6 months after randomization
  TCD is used to evaluate the change in cerebral blood flow (cm/s) 6 months after treatment. Higher speed mean a worse outcome.
The change of middle cerebral artery pulsatility index at 6 months | 3 months and 6 months after randomization
  TCD is used to evaluate the change of middle cerebral artery pulsatility index at 6 months. Higher pulsatility index mean a worse outcome.

SECONDARY OUTCOMES:
cognitive function assessed by MoCA at 6 months | 6 months after randomization
  Cognition function assessed by Montreal Cognitive Assessment (MoCA) score. Score range 0-30. Higher scores mean a better outcome.
cognitive function assessed by Clinical Dementia Rating (CDR) at 6 months | 6 months after randomization
  Cognitive function assessed by Clinical Dementia Rating (CDR). Score range 0-3. Higher scores mean a worse outcome.
The change of White Matter hyperintense volume at 6 months | 6 months after randomization
  WMH volume is assessed on 3D fluid attenuated inversion recovery (FLAIR) sequence in mm3 or cm3. Larger volume indicates a worse outcome.
The change of White Matter hyperintensities Fazekas scores at 6 months | 6 months after randomization
  Fazekas score is used to describe the different types of hyperintense signal abnormalities surrounding the ventricles and in the deep white matter. Periventricular hyperintensity (PVH) is graded as 0 = absence, 1 = "caps" or pencil-thin lining, 2 = smooth "halo", 3 = irregular PVH extending into the deep white matter. Separate deep white matter hyperintensity (DWMH) is rated as 0 = absence, 1 = punctate foci, 2 = beginning confluence of foci, 3 = large confluent areas. Higher scores indicats a worse outcome.
The change of Cerebral blood flow values for MRI cerebral perfusion imaging at 6 months | 6 months after randomization
  MRI is used to evaluate the change of Cerebral blood flow values for MRI cerebral perfusion imaging at 6 months.
Digit span test | 6 months after randomization
  The Digit span test is used to assess cognitive function change for 6 months. The score ranges from 0 to 44. Higher scores mean a better outcome.
Stroop Color Word Test | 6 months after randomization
  The Stroop Color and Word Test is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. Shorter the test time, the better the outcome.
Hamilton Anxiety Scale(HAMA) | 6 months after randomization
  Mood function is assessed by Hamilton Anxiety Scale(HAMA). The Score ranges 0-56. Higher scores mean a worse outcome.
Hamilton Depression Scale(HAMD) | 6 months after randomization
  Mood function assessed by Hamilton Depression Scale(HAMD). The Score ranges 0-68. Higher scores mean a worse outcome.
The Short Physical Performance Battery(SPPB) | 6 months after randomization
  It is a composite measure assessing walking speed, standing balance, and sit-to-stand performance. It has primarily been used to assess elderly patients both in the hospital and community setting.
Urination and defecation | 6 months after randomization
  The score of the urination and defecation function scale changed at 6 months.

OTHER OUTCOMES:
Neurovascular coupling index | 3 months and 6 months after randomization
  Data are presented as peak population normalized mean changes from baseline, and median area under the curve (AUC).
Electroencephalogram oscillations | 3 months and 6 months after randomization
  The amplitude, frequency, phase, coherence will be measured.
Blood-Brain Barrier (BBB) Permeability between groups. | 3 months and 6 months after randomization
  BBB permeability is assessed by MRI and biomarker (including NSE, GFAP, S100β).

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wang, PhD，MD, Principal Investigator — Beijing Tiantan Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Tiantan Hospital, Beijing, China